CLINICAL TRIAL: NCT02395016
Title: A Prospective, Randomized, Controlled, Double-blind, Multi-center Clinical Study of Nimotuzumab Combinated With Gemcitabine Contrast to Placebo Combinated With Gemcitabine in K-RAS Wild-type,Locally Advanced and Metastatic Pancreatic Cancer
Brief Title: A Study of Nimotuzumab Combinated With Gemcitabine in K-RAS Wild-type Locally Advanced and Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Collaborators: NanJing PLA 81 Hospital (Other); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPL-Nim-PC-1
Record Dates: First submitted 2015-01-17; First posted 2015-03-20 (Estimated); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — nimotuzumab; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nimotuzumab and Gemcitabine (Experimental): nimotuzumab,400mg/w，Intravenous infusion over 60 minutes,Until disease progression or intolerable toxicity or subjects ask to leave the test.
  Gemcitabine，1000mg/m2，Intravenous infusion over 30 minutes,Once every three weeks, rest one week (d1,8,15; q28d), Every 4 weeks for a period,Until disease progression or intolerable toxicity or subjects ask to leave the test.
  Interventions: Drug: nimotuzumab; Drug: Gemcitabine
- Placebo and Gemcitabine (Placebo Comparator): placebo,400mg/w，Intravenous infusion over 60 minutes,Until disease progression or intolerable toxicity or subjects ask to leave the test.
  Gemcitabine，1000mg/m2，Intravenous infusion over 30 minutes,Once every three weeks, rest one week (d1,8,15; q28d), Every 4 weeks for a period,Until disease progression or intolerable toxicity or subjects ask to leave the test.
  Interventions: Drug: Gemcitabine; Other: Placebo

INTERVENTIONS:
Drug: nimotuzumab — nimotuzumab,400mg/w，Intravenous infusion over 60 minutes,Until disease progression or intolerable toxicity or subjects ask to leave the test.
  Other Names: Taixinsheng
  Arms: Nimotuzumab and Gemcitabine
Drug: Gemcitabine — Gemcitabine，1000mg/m2，Intravenous infusion over 30 minutes,Once every three weeks, rest one week (d1,8,15; q28d), Every 4 weeks for a period,Until disease progression or intolerable toxicity or subjects ask to leave the test.
Other: Placebo — Placebo，400mg/w，Intravenous infusion over 60 minutes,Until disease progression or intolerable toxicity or subjects ask to leave the test.
  Arms: Placebo and Gemcitabine

SUMMARY:
Nimotuzumab is a humanized monoclonal antibody against epidermal growth factor receptor (EGFR). Clinical trials are ongoing globally to evaluate Nimotuzumab in different indications. Nimotuzumab has been approved to treat squamous cell carcinoma of head and neck (SCCHN), glioma and nasopharyngeal carcinoma in different countries.The clinical phase Ⅲ trial designed to assess overall survival（OS）of the combination of Nimotuzumab administered concurrently with Gemcitabine in patients with RAS wild type of locally advanced or metastatic pancreatic cancer

DETAILED DESCRIPTION:
Nimotuzumab is a humanized monoclonal antibody against epidermal growth factor receptor (EGFR). Clinical trials are ongoing globally to evaluate Nimotuzumab in different indications. Nimotuzumab has been approved to treat squamous cell carcinoma of head and neck (SCCHN), glioma and nasopharyngeal carcinoma in different countries.The clinical phase Ⅲ trial designed to assess overall survival（OS）of the combination of Nimotuzumab administered concurrently with Gemcitabine in patients with RAS wild type of locally advanced or metastatic pancreatic cancer.Secondary objectives include time to progression（TTP）,progression-free survival（PFS）,Objective Response Rate（ORR）,Disease Control Rate（DCR）,Clinical Benefit Response（CBR）and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-75 years old
* KPS≥60
* Histological or cytological diagnosis that are unsuitable for radical radiotherapy or surgical treatment of locally advanced or metastatic pancreatic adenocarcinoma (≥6 months to the last adjuvant chemotherapy)
* Has at least one objective measurable lesion can be evaluated according to Response Evaluation Criteria in Solid Tumors1.1(Helical CT examination of the longest diameter of target lesions≥10mm, such as lymph node metastasis only need the shortest path ≥15mm)
* Life expectancy ≥12 weeks
* K-RAS tumor tissue detected as the wild-type
* Aspartate transaminase（AST）/aminotransferase（ALT）≤2.5×ULN，AST /ALT≤5×ULN（if liver metastases）；Total bilirubin≤2×ULN，Total bilirubin≤3×ULN（if liver metastases）；Absolute neutrophil count≥1.5×109/L；Blood platelet≥100×109/L；Hemoglobin≥90 g/L；Creatinine clearance≥60ml/min
* Volunteered to participate this study, written informed consent and has a good compliance
* Patients of childbearing age and their spouses are willing to take contraceptive measures

Exclusion Criteria:

* Before this study had received the following treatments：As a means of anti-tumor palliative chemotherapy and molecular targeted therapy.Target lesion had received radiotherapy without progression.within 4 weeks or be participating in clinical trials of other therapeutic/ interventionist clinical trial.
* Undergone major surgery within 4 weeks.
* The brain metastasis or leptomeningeal metastasis.
* Has a history of malignancy other than the pancreatic cancer (except for the cured cervix in situ or basal cell carcinoma, and a five-year cure other cancers).
* The merger has symptoms of ascites and requires clinical treatment. Accompanied by other serious disease, including but not limited:Congestive heart failure which is difficult to control (NYHA III or IV), Unstable angina, Poorly controlled arrhythmia, Uncontrolled moderate to severe hypertension(systolic blood pressure（SBP）>160 mm Hg or diastolic blood pressure（DBP）>100 mm Hg).Active infection.Diabetes which is difficult to control.Has mental illness which impacts the informed consent and / or compliance program.HIV infection.There is serious illness that other researchers consider is unsuitable to participate this study.
* Known allergy to anti-EGFR antibody formulations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: shukui qin, MD, PHD, Principal Investigator — 81th Hospital of PLA; jin li, MD, PHD, Principal Investigator — Fudan University
Locations (25):
- China (25):
  - First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Union Medical College Hospital, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality
  - PLA General Hospital (301 Hospital), Beijing, Beijing Municipality
  - Affiliated Hospital of Military Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fuzhou General Hospital of Nanjing Military Region, Fuzhou, Fujian
  - Fujian Provincial Tumor Hospital, Fuzhou, Fujian
  - Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Jiangyin City People's Hospital, Jiangyin, Jiangsu
  - Jiangsu Province Tumor Hospital, Nanjing, Jiangsu
  - Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shanghai Jiaotong University Affiliated Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - First People's Hospital Cancer Center, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Affiliated Xijing Hospital, Fourth Military Medical University, Xi’an, Shanxi
  - General Hospital of Chengdu Military Region, Chengdu, Sichuan
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Qin S, Li J, Bai Y, Wang Z, Chen Z, Xu R, Xu J, Zhang H, Chen J, Yuan Y, Liu T, Yang L, Zhong H, Chen D, Shen L, Hao C, Fu D, Cheng Y, Yang J, Wang Q, Qin B, Pan H, Zhang J, Bai X, Zheng Q. Nimotuzumab Plus Gemcitabine for K-Ras Wild-Type Locally Advanced or Metastatic Pancreatic Cancer. J Clin Oncol. 2023 Nov 20;41(33):5163-5173. doi: 10.1200/JCO.22.02630. Epub 2023 Aug 30. PMID 37647576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We screened 480 patients between April 10, 2015, and September 2020, at 25 study sites in China. Finally, 90 patients with K-Ras gene wild-type were enrolled.
Groups:
- Nimotuzumab and Gemcitabine: nimotuzumab,400mg/w，Intravenous infusion over 60 minutes,Until disease progression or intolerable toxicity or subjects ask to leave the test.
  Gemcitabine，1000mg/m2，Intravenous infusion over 30 minutes,Once every three weeks, rest one week (d1,8,15; q28d), Every 4 weeks for a period,Until disease progression or intolerable toxicity or subjects ask to leave the test.
  nimotuzumab: nimotuzumab,400mg/w，Intravenous infusion over 60 minutes,Until disease progression or intolerable toxicity or subjects ask to leave the test.
  Gemcitabine: Gemcitabine，1000mg/m2，Intravenous infusion over 30 minutes,Once every three weeks, rest one week (d1,8,15; q28d), Every 4 weeks for a period,Until disease progression or intolerable toxicity or subjects ask to leave the test.
- Placebo and Gemcitabine: placebo,400mg/w，Intravenous infusion over 60 minutes,Until disease progression or intolerable toxicity or subjects ask to leave the test.
  Gemcitabine，1000mg/m2，Intravenous infusion over 30 minutes,Once every three weeks, rest one week (d1,8,15; q28d), Every 4 weeks for a period,Until disease progression or intolerable toxicity or subjects ask to leave the test.
  Gemcitabine: Gemcitabine，1000mg/m2，Intravenous infusion over 30 minutes,Once every three weeks, rest one week (d1,8,15; q28d), Every 4 weeks for a period,Until disease progression or intolerable toxicity or subjects ask to leave the test.
  Placebo: Placebo，400mg/w，Intravenous infusion over 60 minutes,Until disease progression or intolerable toxicity or subjects ask to leave the test.
Period: Overall Study
Arm/Group | Nimotuzumab and Gemcitabine | Placebo and Gemcitabine
Started | 45 | 45
Completed | 30 | 33
Not Completed | 15 | 12
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Protocol Violation | 2 | 3

BASELINE CHARACTERISTICS:
Population: We screened 90 pts from 480 pts, of whom 8 pts were excluded due to serious violation of the inclusion criteria: 7 pts with K-Ras mutants, 1 pt with gallbladder cancer. Finally, 82 pts were included in FAS.
Groups:
- Nimotuzumab- Gemcitabine Group: receive nimotuzumab (400 mg, weekly) plus gemcitabine (1000 mg/m2 on days 1, 8, and 15, every four weeks) until disease progression or unacceptable toxicity.
- Placebo-Gemcitabine Group: receive Placebo plus gemcitabine (1000 mg/m2 on days 1, 8, and 15, every four weeks) until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Nimotuzumab- Gemcitabine Group | Placebo-Gemcitabine Group | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 30 | 63
  >=65 years | 8 | 11 | 19
Age, Continuous [Median (Full Range); unit: years] | 53 [19 to 73] | 57 [19 to 73] | 55 [19 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 27 | 24 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han | 41 | 39 | 80
  Others | 0 | 2 | 2
Karnofsky performance-status score [Count of Participants; unit: Participants] — The KPS score ranges from 0 to 100, with a higher score indicating better performance status. The scoring is subjectively assigned by a health professional based on the following hierarchical scale: 100=normal, no evidence of disease; 90=able to perform normal activity with only minor symptoms; 80=normal activity with effort, some symptoms; 70=able to care for self but unable to do normal activities; 60=requires occasional assistance, care for most needs.
  Participants
    90-100 score | 20 | 22 | 42
    60-80 score | 21 | 19 | 40
Diagnosis [Count of Participants; unit: Participants]
  Locally advanced | 9 | 8 | 17
  Metastatic | 32 | 33 | 65
Pancreatic tumor location [Count of Participants; unit: Participants]
  Head | 17 | 17 | 34
  Body | 6 | 7 | 13
  Tail | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival（OS）
Description: The primary endpoint was overall survival (OS, defined as from randomization to death due to any cause).
  We screened 90 pts (90 patients were allocated for treatment) from 480 pts, of whom 8 pts were excluded due to serious violation of the inclusion criteria: 7 pts with K-Ras mutants, 1 pt with gallbladder cancer. Finally, 82 pts were included in FAS. The primary end point was evaluated in the full analysis set (FAS; all eligible patients who received at least one dose of nimotuzumab/placebo and had one evaluation of efficacy).
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Nimotuzumab- Gemcitabine Group: receive nimotuzumab (400 mg, weekly) plus gemcitabine until disease progression or unacceptable toxicity
- Placebo-Gemcitabine Group: receive placebo plus gemcitabine until disease progression or unacceptable toxicity
Arm/Group | Nimotuzumab- Gemcitabine Group | Placebo-Gemcitabine Group
Number analyzed (Participants) | 41 | 41
months | 10.9 [5.6 to 16.3] | 8.5 [5.7 to 10]

2. Secondary Outcome: Time to Progression（TTP）
Description: TTP, defined as from randomization to the first observation of disease progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: up to 3 years
Population: We screened 90 pts (90 patients were allocated for treatment) from 480 pts, of whom 8 pts were excluded due to serious violation of the inclusion criteria: 7 pts with K-Ras mutants, 1 pt with gallbladder cancer. Finally, 82 pts were included in FAS. Secondary end points were analyzed only in the FAS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nimotuzumab- Gemcitabine Group | Placebo-Gemcitabine Group
Number analyzed (Participants) | 41 | 41
months | 4.7 [2.7 to 9] | 3.7 [2 to 5.4]

3. Secondary Outcome: Progression Free Survival（PFS）
Description: PFS, defined as from randomization to disease progression or all-cause death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: up to 3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nimotuzumab- Gemcitabine Group | Placebo-Gemcitabine Group
Number analyzed (Participants) | 41 | 41
months | 4.2 [2.7 to 7.3] | 3.6 [2 to 5]

4. Secondary Outcome: Objective Response Rate（ORR）
Description: Objective response rate (ORR), including complete response (CR) and partial response (PR). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Once every eight weeks，up to 5.4 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimotuzumab- Gemcitabine Group | Placebo-Gemcitabine Group
Number analyzed (Participants) | 41 | 41
Participants | 3 | 4

5. Secondary Outcome: Disease Control Rate（DCR）
Description: Disease control rate (DCR), including complete response (CR) and partial response (PR) and stable disease(SD). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: CR, disappearance of all target lesions; PR, at least a 30% decrease in the sum of the longest diameter of target lesions. SD, neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (PD, defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions).
Time Frame: Once every eight weeks，up to 5.4 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Nimotuzumab- Gemcitabine Group | Placebo-Gemcitabine Group
Number analyzed (Participants) | 41 | 41
Participants | 28 | 26

6. Secondary Outcome: Clinical Benefit Response（CBR）
Description: The clinical benefit response(CBR)was evaluated every 8 weeks on the basis of the Burris criteria. CBR included pain (intensity of pain and consumption of analgesics), PS (performance status, evaluated according to KPS) and weight changes. Effective is defined as at least one positive improvement in the CBR index (pain, physical status or weight change) and no negative indicator is found, which can be rated as a clinical benefit case.
Time Frame: every 8 weeks, up to 5.4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Nimotuzumab- Gemcitabine Group | Placebo-Gemcitabine Group
Number analyzed (Participants) | 28 | 31
Participants | 11 | 10

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse Events as any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Time Frame: up to 75.2 months
Population: We screened 90 pts from 480 pts, of whom 8 pts were excluded due to serious violation of the inclusion criteria: 7 pts with K-Ras mutants, 1 pt with gallbladder cancer. Finally, 90 pts were included in SS (safety set). Adverse Events were analyzed in the SS (n=90).
Measure: Number; unit: participants
Arm/Group | Nimotuzumab- Gemcitabine Group | Placebo-Gemcitabine Group
Number analyzed (Participants) | 45 | 45
participants
  Treatment-related Adverse Events | 31 | 29
  Serious Adverse Events | 1 | 2
  Drug reduction or discontinued for AE | 4 | 6
  Withdrawal for AE | 2 | 1
  All-Cause Mortality | 36 | 40

ADVERSE EVENTS:
Time Frame: up to 75.2 months
Description: We screened 90 pts from 480 pts, of whom 8 pts were excluded due to serious violation of the inclusion criteria: 7 pts with K-Ras mutants, 1 pt with gallbladder cancer. Finally, 90 pts were included in SS (safety set). Adverse Events were analyzed in the SS.
Arm/Group | Nimotuzumab- Gemcitabine Group | Placebo-Gemcitabine Group
All-Cause Mortality (participants affected / at risk) | 36/45 | 40/45
Serious Adverse Events (participants affected / at risk) | 15/45 | 5/45
Other Adverse Events (participants affected / at risk) | 44/45 | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimotuzumab- Gemcitabine Group (N=45) | Placebo-Gemcitabine Group (N=45)
Fever (General disorders) | 1 | 0
ileus (Gastrointestinal disorders) | 1 | 0
enteritis (Gastrointestinal disorders) | 0 | 1
stomachache (Gastrointestinal disorders) | 1 | 0
vomiting (Gastrointestinal disorders) | 0 | 1
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
bilirubin increased (Investigations) | 2 | 0
weight decreased (Investigations) | 0 | 1
Hemoglobin decreased (Investigations) | 1 | 0
platelet count decreased (Investigations) | 1 | 0
Embolic cerebral infarction (Vascular disorders) | 1 | 0
diabetic neuropathy (Nervous system disorders) | 1 | 0
coagulopathy (Blood and lymphatic system disorders) | 2 | 0
anemia (Blood and lymphatic system disorders) | 1 | 0
hypoproteinemia (Metabolism and nutrition disorders) | 1 | 0
cholecystitis (Hepatobiliary disorders) | 1 | 0
tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimotuzumab- Gemcitabine Group (N=45) | Placebo-Gemcitabine Group (N=45)
white blood cell count decreased (Investigations) | 34 | 26
utrophil count decreased (Investigations) | 31 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-06-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT02395016/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT02395016/SAP_001.pdf